CLINICAL TRIAL: NCT03622151
Title: Homeless Population and Mental Health: Impact of Primer la Llar Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Sanitari Sant Joan de Déu (Other)
Responsible Party: Principal Investigator, Inés Campo Ferreiro, Mental Health Nurse, Parc Sanitari Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PIC-130-15
Record Dates: First submitted 2018-07-18; First posted 2018-08-09 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Mental Health Disorder
Keywords: mental health; Housing First; homeless
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Intervention group (housing first model program) and control group (treatment as usual).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Primer la Llar Program (housing first model): to live in permanent and individual housing and receiving weekly visits from a multidisciplinary team.
  Interventions: Other: Primer la Llar program
- Control group (No Intervention): Treatment as usual:
  attention from the resources of the homeless network in Barcelona.

INTERVENTIONS:
Other: Primer la Llar program — Housing First model: permanent housing without previous requirements such as abstinence, sobriety or compliance with treatment.
  Arms: Intervention group

SUMMARY:
The main goal is to evaluate the impact of the Primer La Llar housing program for the homeless population on the mental health of the participants.

The hypothesis is that the housing program, which follows Housing first model, for the homeless population has a positive impact on the mental health of the participants, compared to the group that does not receive the intervention -treatment as usual group (meaning the "positive impact" a lower score on the symptomatology scales and lower toxic intake in the group receiving the intervention).

DETAILED DESCRIPTION:
The specific objectives are:

Identify the socio-demographic and clinical characteristics of the participants.

Compare the severity of psychiatric symptoms and improvement among the participants in the intervention group and the control group (depressive, anxious, psychotic or manic symptomatology, depending on the case).

Compare the consumption of alcohol and drugs among the participants of both groups.

Compare the basic daily life skills among the participants in both groups, as well as the improvement of them in the experimental group.

Compare the use of services and between the participants of the intervention group and the control group.

Intervention group receives entry to the program (which means individual and permanent housing without previous requirements such as abstinence, compliance with treatment or sobriety.

Control group receives treatment as usual, as they are users of homeless population network of Barcelona.

ELIGIBILITY:
Inclusion Criteria:

* Single people, adults (exceptionally sentimental couples, friends with positive support relationship for both).
* Long life on the street (minimum 1 year staying overnight on the street) and / or accommodation centers without linking, using them in a timely manner in the last year.
* Social needs concurrent to the lack of housing: mental illness and / or drug abuse.
* Functional autonomy for daily life.
* Have regular economic income or possibility of obtaining them.
* Sign informed consent form.

Exclusion Criteria:

* language barrier
* severe neurological or organic pathology
* severe dementia
* alcoholic dementia Wernicke Korsakoff

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Prevalence and gravity of psychotic symptoms in both groups | Up to 21 months
  PANSS scale (Positive And Negative Syndrome Scale). Subscales: 1. PANSS-P-Positive (7 ítems): range 7-49 (minimum and maximum scores) 2. PANSS-N-Negative (7 ítems). Range: 7-49. 3. PANSS-PG- general psychopathology (16 ítems). Range: 16-112. Higher values represent a worse outcome. Subscales are summed to compute a total score.
Prevalence and gravity of anxious symptoms in both groups | Up to 21 months
  HARS scale (Hamilton Anxiety Rating Scale). Total range:0-56. Higher values represent a worse outcome.
Prevalence and gravity of depressive symptoms in both groups | Up to 21 months.
  HDRS scale (Hamilton Depression Rating Scale). Total range: 0-52. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Changes in number of visits to the emergency room/health center/specialist doctors | Up to 21 months
  To see if there are increases or decreases in use of general and specific health services; questionnaire on use of services.
Basic skills of daily life | Up to 21 months
  BELS scale (Basic everyday living skills). Range subscales:
  self-care (0-40) domestic skills (0-28) community skills (0-16) and activity and social relations (0-20). Higher value reports better outcome. Subescales are summed to compute a total score.
Sociodemographic and psychopathological description of both groups | Up to 21 months
  Number of participants from each country, average age, number of men and women, number of participants with a problem of substance abuse or mental health, etc.
  Assessed by a questionnaire about clinical and socio-demographic items.
Number of participants with an alcohol abuse problem assessed by Audit test | Up to 21 months
  Changes in alcohol abuse in both groups Audit test (0-40). Higher value reports worse outcome.
Number of participants with a drug abuse problem assessed by questionnaire on drug abuse | Up to 21 months
  Increase or decrease on drug abuse in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Haro Abad, Study Director — Parc Sanitari Sant Joan de Déu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aubry T, Tsemberis S, Adair CE, Veldhuizen S, Streiner D, Latimer E, Sareen J, Patterson M, McGarvey K, Kopp B, Hume C, Goering P. One-year outcomes of a randomized controlled trial of housing first with ACT in five Canadian cities. Psychiatr Serv. 2015 May 1;66(5):463-9. doi: 10.1176/appi.ps.201400167. Epub 2015 Feb 2. PMID 25639993
- [Background] Henwood BF, Byrne T, Scriber B. Examining mortality among formerly homeless adults enrolled in Housing First: An observational study. BMC Public Health. 2015 Dec 4;15:1209. doi: 10.1186/s12889-015-2552-1. PMID 26634243
- [Background] Kerman N, Sylvestre J, Aubry T, Distasio J. The effects of housing stability on service use among homeless adults with mental illness in a randomized controlled trial of housing first. BMC Health Serv Res. 2018 Mar 20;18(1):190. doi: 10.1186/s12913-018-3028-7. PMID 29558927
- [Background] Somers JM, Patterson ML, Moniruzzaman A, Currie L, Rezansoff SN, Palepu A, Fryer K. Vancouver At Home: pragmatic randomized trials investigating Housing First for homeless and mentally ill adults. Trials. 2013 Nov 1;14:365. doi: 10.1186/1745-6215-14-365. PMID 24176253
- [Background] Stergiopoulos V, Hwang SW, Gozdzik A, Nisenbaum R, Latimer E, Rabouin D, Adair CE, Bourque J, Connelly J, Frankish J, Katz LY, Mason K, Misir V, O'Brien K, Sareen J, Schutz CG, Singer A, Streiner DL, Vasiliadis HM, Goering PN; At Home/Chez Soi Investigators. Effect of scattered-site housing using rent supplements and intensive case management on housing stability among homeless adults with mental illness: a randomized trial. JAMA. 2015 Mar 3;313(9):905-15. doi: 10.1001/jama.2015.1163. PMID 25734732